CLINICAL TRIAL: NCT06503263
Title: Zanubrutinib and Lenalidomide as Maintenance Therapy in Patients With Diffuse Large B-cell Lymphoma
Brief Title: Zanubrutinib and Lenalidomide as Maintenance Therapy in DLBCL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Navy General Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Liren Qian, Vice Director, Navy General Hospital, Beijing
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZLDLBCL2024
Record Dates: First submitted 2024-07-10; First posted 2024-07-16 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Diffuse Large B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — zanubrutinib; Lenalidomide; Maintenance

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maintenance Therapy (Experimental): Patients were treated by Zanubrutinib plus Lenalidomide as Maintenance Therapy
  Interventions: Drug: Zanubrutinib plus Lenalidomide as Maintenance Therapy
- No maintenance Therapy (No Intervention): Patients received no maintenance Therapy

INTERVENTIONS:
Drug: Zanubrutinib plus Lenalidomide as Maintenance Therapy — Patients were treated by Zanubrutinib(160mg po bid d1-28) plus Lenalidomide(25mg po qd d1-14) as maintenance therapy until 2 years post chemotherpay
  Other Names: Zanubrutinib plus Lenalidomide
  Arms: Maintenance Therapy

SUMMARY:
The goal of this phase 2 trial is to test the safety and efficacy of zanubrutinib and lenalidomide as maintenance therapy in patients with DLBCL.

DETAILED DESCRIPTION:
The investigators will evaluate safety and efficacy of zanubrutinib and lenalidomide as maintenance therapy in patients with diffuse large B-cell lymphoma post complete remission and have completed planed courses of chemotherapy . Event-free survival (EFS), progression-free survival (PFS), overall survival (OS), adverse events (AEs) will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed Diffuse Large B Cell Lymphoma according World Health Organization (WHO) classification;
* Patient is ≥ 18 years of age at the time of signing the informed consent form (ICF).
* Patient must understand and voluntarily sign an ICF prior to any study-specific assessments/procedures being conducted;
* Patient is willing and able to adhere to the study visit schedule and other protocol requirements;
* Patient has recieved complete remission and has completed planed courses of chemotherapy
* Meet the following lab criteria: Absolute Neutrophil Count (ANC) ≥ 1,5 x 10^9/L (≥ 1 x 10^9/L if bone marrow (BM) involvement by lymphoma)；Platelet ≥ 75 x 10^9/L (≥ 50 x 10^9/L if BM involvement by lymphoma)； Hemoglobin ≥ 8 g/dL. Anticipated life expectancy at least 3 months

Exclusion Criteria:

* Active or uncontrolled infections requiring systemic treatment within 14 days before enrollment;
* Any instability of systemic disease, including but not limited to severe cardiac, liver, kidney, or metabolic disease need therapy;
* Pregnant or lactating women

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-08-30 (Actual); Primary Completion 2030-07-30 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
EFS | 2 years
  EFS was defined as the time from treatment initiation to progression, relapse, new treatment, or death by any cause, whichever occurred first.

SECONDARY OUTCOMES:
PFS | 2 years
  PFS was defined as the time from study entry until disease progression or death by any cause
OS | 2 years
  OS was defined as the time from treatment initiation to death by any cause.

CONTACTS AND LOCATIONS:
Overall Officials: qlr2007@126.com Qian, PhD, Principal Investigator — Navy General Hospital, Beijing
Locations (1):
- Navy General Hospital, Beijing, Beijing Municipality, China